CLINICAL TRIAL: NCT07306065
Title: Scientific Proof of Music Therapy's Impact on Alzheimer's Disease
Brief Title: University of Central Florida Music Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007771
Record Dates: First submitted 2025-10-08; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Alzheimers Disease; Dementia; Dementia Alzheimer Type
Keywords: Alzheimer s disease; music; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: The study intervention is music, which is being provided by a UCF music concert where the participants will listen to symphonic music.
Masking Description: All participants will undergo the same intervention. Each participant will be assigned a participant ID. All research data will be associated with the participant ID only and not with any of the participant's personal identifiers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants in study will undergo music intervention.
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — UCF music concert where the participants will listen to symphonic, classical music for 1 hour.

SUMMARY:
The purpose of this study is to scientifically validate the impact of music therapy on Alzheimer's disease (AD) by analyzing molecular biomarkers in salivary exosomes. Exosomes are extracellular vesicles that carry molecular signals from brain cells, providing a non-invasive method to assess physiological changes.

DETAILED DESCRIPTION:
Music therapy has long been recognized as a beneficial intervention for individuals with Alzheimer's disease (AD), with evidence supporting improvements in mood, cognitive function, and behavioral symptoms. However, despite widespread clinical use, the biological mechanisms underlying these benefits remain poorly understood. Most studies on music therapy in AD have relied on behavioral observations and qualitative assessments, lacking objective, molecular-level validation. Recent advancements in exosome research have opened new possibilities for non-invasive biomarker analysis. Exosomes, small extracellular vesicles released by cells, carry molecular signatures that reflect physiological states, including neurochemical changes associated with AD.

However, to date, no study has investigated whether music therapy induces measurable changes in exosome biomarkers related to AD pathology.

Key gaps in current knowledge include:

1. Lack of molecular validation for music therapy: While clinical benefits have been reported, no study has demonstrated the neurochemical effects of music therapy on biomolecular markers.
2. Unclear mechanisms of action: It remains unknown whether music therapy modulates neurotransmitter levels (serotonin, dopamine) or pathological proteins (amyloid-beta, tau) associated with AD.
3. Absence of personalized treatment approaches: Without biomarker-based validation, music therapy is typically applied in a one-size-fits-all manner, rather than being tailored to individual neurochemical profiles.
4. Limited non-invasive monitoring tools: Current methods for assessing treatment efficacy rely on neuroimaging or invasive procedures, which are costly and impractical for routine clinical use.

This study seeks to address these gaps by leveraging salivary exosomes as a novel, non-invasive platform to quantify molecular changes induced by music therapy in AD patients.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old or older.

  * 20 adults with no mild-cognitive impairment
  * 20 adults with mild-cognitive impairment
  * 20 adults with Alzheimer's disease/ dementia.
* participant or the participant's legally authorized representative must be able to read or speak English and agree to comply with study procedures.
* pregnant women may chose to participate

Exclusion Criteria:

* 49 years and younger
* prisoners
* unable to understand English and provide consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Effect of music therapy in Alzheimer's patients by analyzing salivary exosomes | 6 months
  To determine the effect of music therapy on key neurochemical biomarkers in Alzheimer's patients by analyzing serotonin, dopamine, amyloid-beta, and tau protein levels in salivary exosomes before and after music therapy sessions.

SECONDARY OUTCOMES:
Identifying therapeutic benefits by correlating changes in biomarkers | 6 months
  To establish a molecular basis for the therapeutic benefits of music therapy by correlating changes in biomarker levels with cognitive, emotional, and behavioral outcomes in AD patients.
Identify differences in individual participant biomarkers | 6 months
  To explore the potential for personalized music therapy by identifying individual differences in biomarker responses, which could guide tailored therapeutic interventions for optimal patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kiminobu Sugaya, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States